CLINICAL TRIAL: NCT04356963
Title: Adjunct Virtual Reality Pain Management in Acute Brain Injury
Brief Title: Adjunct VR Pain Management in Acute Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Nicholas Morris, Assistant Professor of Neurology, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP - 00090603; 1UL1TR003098 (NIH)
Record Dates: First submitted 2020-04-19; First posted 2020-04-22 (Actual); Results first posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Traumatic Brain Injury; Headaches Posttraumatic; Trauma; Pain, Acute
MeSH Terms: conditions — Brain Injuries, Traumatic; Post-Traumatic Headache; Wounds and Injuries; Acute Pain

STUDY DESIGN:
Intervention Model Description: Within-Subjects Design. All participants (single group, 1 arm) intended to complete all three sessions (interventions) in randomized order. At least 4 hours were required to pass between each session to allow for washout.
Masking Description: Interventions will take place in patient rooms with curtain pulled and sign to mask active intervention vs. control intervention from care providers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Experimental): All patients were intended to engage in three different 20-30 min sessions run by research coordinators and spaced a minimum of 4 hours apart to allow for washout of effects, including 1) a commercially available, immersive VR environment, theBlu (WEVR, Inc, Venice, California, USA) delivered via Oculus Rift (Oculus VR, Irvine, California, USA) headset (VR Blu), 2) a non-immersive two-dimensional mimic delivered via a tablet computer (Tablet Blu), and 3) a VR control session delivered via a content-less Oculus Rift headset (VR Blank). The three sessions were run by research coordinators and spaced a minimum of 4 hours apart. The intervention order was counterbalanced using a randomized sequence generator.
  Interventions: Behavioral: Virtual Reality Session (VR Blu); Behavioral: Tablet-based Session (Tablet Blu); Behavioral: Use of Virtual Reality Head Mounted Display without Content (VR Blank)

INTERVENTIONS:
Behavioral: Virtual Reality Session (VR Blu) — 20-30 minute session of virtual reality immersive content.
Behavioral: Tablet-based Session (Tablet Blu) — 20-30 minute session of tablet-based content that mimics the content from virtual reality sessions.
Behavioral: Use of Virtual Reality Head Mounted Display without Content (VR Blank) — 20-30 minutes session using head mounted display to reduce light and sound.

SUMMARY:
Severe and refractory pain after acute injury is a known-risk factor for chronic opioid use disorder. In this study, the investigators will use Virtual Reality (VR) immersion as a non-pharmacological adjunct to treat pain associated with acute traumatic injuries, including traumatic brain injury. The investigators hypothesize that VR therapy will decrease pain and reduce opioid use in patients with acute traumatic injuries, including TBI.

DETAILED DESCRIPTION:
Each participant will undergo one VR session and two control sessions. The VR session will take place in a commercially available VR environment, the Blu, and last 20-30 minutes (VR Blu). The control sessions will include a 2D-tablet based session that mimics the VR content (Tablet Blu) and a content-less placement of the VR headset (VR Blank). The order of these sessions will be randomized across participants are intended to complete all sessions.

Each participant will complete a pre-study questionnaire to elicit their prior experience with the virtual reality as well as measures of gaming addiction/engagement, boredom, and expectancy. These scales will help us determine which patient-level factors predict response to VR. Before and after each session, participants will complete validated scales of pain, nausea, and anxiety.. Pre- and Post-VR opioid use will be recorded. Basic vital signs including heart rate, blood pressure, and respiratory rate, will be recorded before and after each session to monitor autonomic response. Advanced measures of autonomic response will include heart rate variability,,and pupillometry metrics. At the conclusion of all sessions, participants will complete another questionnaire to document their subjective experience of using VR (perceived effectiveness)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Traumatic Injury (including but not limited to traumatic brain injury)
* Age greater than or equal to 18 years-old
* Endorsing at least moderate pain as defined by documentation of at least one numeric rating pain scale score of 3 or more in the last 24 hours.
* Glasgow Coma Scale of 15
* Expected to stay in the hospital for at least 12 hours after enrollment

Exclusion Criteria:

* Seizure prior to enrollment
* Pregnancy
* non-English speaking
* Known intolerance of Virtual Reality
* Patient unable to consent for themselves

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-05 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2022-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas A Morris, M.D., Principal Investigator — University of Maryland, Baltimore
Locations (2):
- United States (2):
  - R Adams Cowley Shock Trauma Center, Baltimore, Maryland
  - University of Maryland Medical Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morris NA, Wang Y, Felix RB, Rao A, Arnold S, Khalid M, Armahizer MJ, Murthi SB, Colloca L. Adjunctive virtual reality pain relief after traumatic injury: a proof-of-concept within-person randomized trial. Pain. 2023 Sep 1;164(9):2122-2129. doi: 10.1097/j.pain.0000000000002914. Epub 2023 Apr 19. PMID 37079851
- [Derived] Felix RB, Rao A, Khalid M, Wang Y, Colloca L, Murthi SB, Morris NA. Adjunctive virtual reality pain relief following traumatic injury: protocol for a randomised within-subjects clinical trial. BMJ Open. 2021 Nov 30;11(11):e056030. doi: 10.1136/bmjopen-2021-056030. PMID 34848527

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2083 patients were screened for eligibility between October 2020 and January 2022 in a dedicated trauma hospital. 1885 patients were excluded. 138 patients declined to participate in the study. 60 patients were enrolled in the study. All patients were intended to participate in all conditions (in randomized order) including: VR Blu, Tablet Blu, VR Blank.
Pre-assignment Details: All 60 patients were intended to participate in all 3 conditions in randomized order. 60 of 60 patients had session order randomized.
Groups:
- All Patients: Patients engaged in three different 20 min sessions run by research coordinators and spaced a minimum of 4 hours apart, including 1) a commercially available, immersive VR environment, theBlu (WEVR, Inc, Venice, California, USA) delivered via Oculus Rift (Oculus VR, Irvine, California, USA) headset (VR Blu), 2) a non-immersive two-dimensional mimic delivered via a tablet computer (Tablet Blu), and 3) a VR control session delivered via a content-less Oculus Rift headset (VR Blank). The three sessions were run by research coordinators and spaced a minimum of 4 hours apart. The intervention order was counterbalanced using a randomized sequence generator. All participants were expected to complete all three sessions.
Period: First Session
Arm/Group | All Patients
Started | 60
Completed VR Blu | 21
Completed Tablet Blu | 19
Completed VR Blank | 19
Completed | 59
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Second Session
Arm/Group | All Patients
Started | 59
Completed VR Blu | 17
Completed Tablet Blu | 23
Completed VR Blank | 15
Completed | 55
Not Completed | 4
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 1
Period: Third Session
Arm/Group | All Patients
Started | 55
Completed VR Blu | 14
Completed Tablet Blu | 12
Completed VR Blank | 22
Completed | 48
Not Completed | 7
Not completed — Lost to Follow-up | 6
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- All Patients: Patients engaged in three different 20 min sessions run by research coordinators and spaced a minimum of 4 hours apart, including 1) a commercially available, immersive VR environment, theBlu (WEVR, Inc, Venice, California, USA) delivered via Oculus Rift (Oculus VR, Irvine, California, USA) headset, 2) a non-immersive two-dimensional mimic delivered via a tablet computer, and 3) a VR control session delivered via a content-less Oculus Rift headset. The three sessions were run by research coordinators and spaced a minimum of 4 hours apart. The intervention order was counterbalanced using a randomized sequence generator.
Arm/Group | All Patients
Number analyzed (Participants) | 60
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53 [38 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 19
  White | 37
  More than one race | 0
  Unknown or Not Reported | 1
Acute Injury Scale > 0 [Number; unit: participants]
  Head | 29
  Head with Traumatic Brain Injury | 20
  Face | 20
  Neck | 8
  Thoracic | 26
  Abdominal | 29
  Spine | 15
  Upper Extremity | 28
  Lower Extremity | 35
Type of Traumatic Brain Injury [Number; unit: participants]
  Intracerebral Hemorrhage | 13
  Subdural hematoma | 10
  Subarachnoid hemorrhage | 8
  Epidural hematoma | 1
Past Medical History [Number; unit: participants]
  Depression | 18
  Anxiety | 16
  Chronic Pain | 13
  Alcohol Abuse | 13
  Positive Toxicology Screen | 32
Health Insurance [Count of Participants; unit: Participants]
  Private | 39
  Medicare | 16
  Medicaid | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Score
Description: Pre- vs. Post-Intervention Ratings on Numeric Pain Rating Scale. Numeric Pain Rating scale range is from 0 (no pain) -10 (severe pain)
Time Frame: Pre- and Post-Intervention (approximately 30 minutes)
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- All Patients: Patients engaged in three different 20 min sessions run by research coordinators and spaced a minimum of 4 hours apart, including 1) a commercially available, immersive VR environment, theBlu (WEVR, Inc, Venice, California, USA) delivered via Oculus Rift (Oculus VR, Irvine, California, USA) headset, 2) a non-immersive two-dimensional mimic delivered via a tablet computer, and 3) a VR control session delivered via a content-less Oculus Rift headset. The three sessions were run by research coordinators and spaced a minimum of 4 hours apart. The intervention order was counterbalanced using a randomized sequence generator.
  Virtual Reality Session: 20-30 minute session of virtual reality immersive content.
  Tablet-based Session: 20-30 minute session of tablet-based content that mimics the content from virtual reality sessions.
  Use of Virtual Reality Head Mounted Display without Content: 20-30 minutes session using head mounted display to reduce light and sound.
Arm/Group | All Patients
Number analyzed (Participants) | 59
score on a scale
  VR Blu Intervention Pain Reduction | -0.92 (0.33)
  Tablet Blu Intervention Pain Reduction | -0.16 (0.29)
  VR Blank Intervention Pain Reduction | -1.24 (0.33)

2. Secondary Outcome: Opioid Administration
Description: Change in amount of opioids received in the 4 hours post-intervention vs. the 4 hours pre-intervention in morphine equivalents
Time Frame: 4 hours post-intervention vs. 4 hours pre-intervention
Measure: Mean (Standard Error); unit: morphine milligram equivalents
Groups:
- All Patients: All patients
Arm/Group | All Patients
Number analyzed (Participants) | 59
morphine milligram equivalents
  Changes in opioid dose received after VR Blu condition | -0.159 (1.392)
  Change in opioid dose received after Tablet Blu | -0.89 (1.175)
  Change in opioid dose received after VR Blank | -0.059 (1.341)

3. Other Pre Specified Outcome: Change in Nausea
Description: Pre- vs. Post-Intervention Ratings on Numeric Rating Scale for Nausea. Numeric Rating Scale for Nausea ranges from 0 (no nausea) - 10 (worst nausea possible)
Time Frame: Pre- and Post-Intervention (approximately 30 minutes)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | All Patients
Number analyzed (Participants) | 59
score on a scale
  Change in nausea after VR Blu | -0.116 (0.304)
  Change in nausea after Tablet Blu | -0.395 (0.248)
  Change in nausea after VR Blank | -0.093 (0.057)

4. Other Pre Specified Outcome: Change in Anxiety
Description: Pre- vs. Post-Intervention Anxiety Ratings from Short-Form State Anxiety Inventory. Scores Range from 6 (Not at all anxious) - 24 (Very much amxious)
Time Frame: Pre- and Post-Intervention (approximately 30 minutes)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | All Patients
Number analyzed (Participants) | 59
score on a scale
  changes in STAI score after VR Blue | -.061 (0.311)
  Changes in STAI score after Tablet Blue | -0.401 (0.32)
  Changes in STAI score after VR Blank | -0.675 (0.501)

5. Other Pre Specified Outcome: Change Heart Rate Variability
Description: Pre- vs. Post-Intervention Heart Rate Variability as measured by normal-to-normal (NN) means. Decreasing NN means are associated with the activity of sympathetic system, while increasing NN means means are associated with the activity of parasympathetic nervous system
Time Frame: Mean NN from last 15 minutes of each intervention compared to mean NN from 15 minutes immediately prior to intervention
Measure: Mean (Standard Error); unit: ms
Arm/Group | All Patients
Number analyzed (Participants) | 25
ms
  VR Blu induced change in mean NN (NN from last 15 min of session minus NN 15 min pre-session) | 874.64 (15.36)
  Tablet Blu induced change in mean NN (NN from last 15 min of session minus NN 15 min pre-session) | 834.78 (1.93)
  VR Blank induced change in mean NN (NN from last 15 min of session minus NN 15 min pre-session) | 867.64 (10.37)

6. Other Pre Specified Outcome: Change in Pupillometry
Description: Pre- vs. Post-Intervention Pupillary Maximum Constriction Velocity. Reduced pupillary maximum constriction velocity is representative of decreased parasympathetic nervous system activity.
Time Frame: Pre- and Post-Intervention (approximately 30 minutes)
Measure: Mean (Standard Error); unit: mm/s
Arm/Group | All Patients
Number analyzed (Participants) | 42
mm/s
  VR Blue change in maximum constriction velocity | 0.187 (0.112)
  Tablet Blue change in maximum constriction velocity | -0.047 (0.097)
  VR Blank change in maximum constriction velocity | -0.299 (0.149)

7. Other Pre Specified Outcome: Subjective Measures of VR Experience
Description: A Likert-Scale questionnaire was used to assess participant's subjective ratings of how effective the interventional sessions were. The scale ranged from 0 (not at all) to 5 (very much).
Time Frame: Pre- and Post-study (approximately 2-3 days)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | All Patients
Number analyzed (Participants) | 59
score on a scale
  VR Blu Perceived Effectiveness on Likert Scale (0-5, not at all effective - very effective) | 3.63 (0.23)
  Tablet Blu Perceived Effectiveness on Likert Scale (0-5, not at all effective - very effective) | 2.68 (0.23)
  VR Blank Perceived Effectiveness on Likert Scale (0-5, not at all effective - very effective) | 1.52 (0.29)

ADVERSE EVENTS:
Time Frame: Duration of Study Involvement (typically < 48 hours)
Description: Potential side-effects of VR were measured before and after each session, including neck pain, nausea, dizziness, and light sensitivity according to a NRS ranging from 0 (no symptom) to 10 (worst possible symptom). Before and immediately after each session, we also collected vital sign measurements (blood pressure and heart rate).
  All participants were intended to participate in all three interventions therefore they are reported as a single arm/group.
Groups:
- All Participants: All Participants were intended to participate in all three interventions.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/54
Serious Adverse Events (participants affected / at risk) | 0/54
Other Adverse Events (participants affected / at risk) | 0/54

LIMITATIONS AND CAVEATS:
Very few patients with TBI met inclusion criteria. The intervals between conditions were quite short to improve feasibility of study completion based on brief anticipated length of stay. This limited our ability to evaluate effects on opioid use and duration of VR intervention effect. The sample size limited our ability to account for multiple comparisons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/63/NCT04356963/Prot_SAP_001.pdf
  • Informed Consent Form (2021-04-15): https://cdn.clinicaltrials.gov/large-docs/63/NCT04356963/ICF_000.pdf